CLINICAL TRIAL: NCT03717415
Title: An Open Label, Multicenter, Phase 1b/2 Study of Rebastinib (DCC-2036) in Combination With Carboplatin to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of Rebastinib (DCC-2036) in Combination With Carboplatin in Patients With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development program terminated.
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2036-01-004
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumor
Keywords: rebastinib; breast cancer; ovarian cancer; mesothelioma
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Ovarian Neoplasms; Mesothelioma | interventions — rebastinib; DCC-2036; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 (Experimental): Dose escalation with rebastinib 50 milligram (mg) twice daily (BID) orally (PO) in 21-day cycles in combination with carboplatin administered by intravenous (IV) infusion at area under the curve (AUC)5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 (Experimental): Dose escalation with rebastinib 100 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 (Experimental): Dose escalation with rebastinib 100 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC6 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 (Experimental): Dose expansion in triple-negative breast cancer (TNBC) participants. Rebastinib 50 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 (Experimental): Dose expansion in TNBC participants. Rebastinib 100 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 (Experimental): Dose expansion in platinum-sensitive ovarian cancer participants. Rebastinib 50 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 (Experimental): Dose expansion in platinum-sensitive ovarian cancer participants. Rebastinib 100 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 (Experimental): Dose expansion in mesothelioma participants. Rebastinib 50 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin
- Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5 (Experimental): Dose expansion in mesothelioma participants. Rebastinib 100 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
  Interventions: Drug: Rebastinib; Drug: Carboplatin

INTERVENTIONS:
Drug: Rebastinib — Administered orally
  Other Names: DCC-2036
Drug: Carboplatin — Administered by IV infusion

SUMMARY:
This is an open-label Phase 1b/2 multicenter study of rebastinib (DCC-2036) in combination with carboplatin designed to evaluate the safety, tolerability, and pharmacokinetics (PK) in participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age at the time of informed consent.
2. Part 1 (Dose Escalation). Histologically confirmed diagnosis of a locally advanced or metastatic solid tumor for which carboplatin is considered appropriate treatment.
3. Part 2 (Dose Expansion)

   * Previously treated, triple-negative breast cancer.
   * Recurrent platinum-sensitive ovarian cancer.
   * Histologically confirmed pleural or peritoneal malignant mesothelioma.
4. ECOG performance status of ≤2.
5. Able to provide an archival tumor tissue sample.
6. Adequate organ function and bone marrow reserve.
7. If a female of childbearing potential, must have a negative pregnancy test prior to enrollment.
8. Patient must provide signed consent to participate in the study and is willing to comply with study-specific procedures.

Exclusion Criteria:

1. Received prior anticancer or other investigational therapy within 28 days or 5× the half-life (whichever is shorter) prior to the first dose.
2. Not recovered from prior-treatment toxicities to Grade ≤1 or baseline.
3. Peripheral neuropathy of any etiology >Grade 1.
4. Concurrent malignancy.
5. Known active CNS metastases.
6. Use of systemic corticosteroids.
7. Known retinal neovascularization, macular edema or macular degeneration.
8. History or presence of clinically relevant cardiovascular abnormalities.
9. QTcF >450 ms in males or >470 ms in females.
10. Left ventricular ejection fraction (LVEF) <50% at screening.
11. Arterial thrombotic or embolic events.
12. Symptomatic venous thrombotic event.
13. Active infection ≥Grade 3.
14. Known HIV or HCV infection only if taking medications excluded per protocol, active HBV, or active HCV infection.
15. Use of proton pump inhibitors.
16. If female, the patient is pregnant or lactating.
17. Major surgery 4 weeks prior to the first dose of study drug.
18. Malabsorption syndrome or other illness which could affect oral absorption.
19. Known allergy or hypersensitivity to any component of rebastinib or any of its excipients.
20. Any other clinically significant comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California San Francisco (UCSF), San Francisco, California
  - UCLA Medical Center, Santa Monica, California
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Started | 3 | 14 | 5 | 9 | 2 | 18 | 2 | 6 | 11
mITT Population (Modified Intent-to-Treat (mITT) Population includes all participants who had at least one full dose of the combined study drugs, had measurable disease at baseline, and had at least one post-baseline assessment. Participants without a post-baseline assessment who discontinued study treatment due to clinical progression, death, or a rebastinib-related AE will also be included in the mITT population.) | 3 | 12 | 5 | 9 | 2 | 18 | 2 | 6 | 11
Completed | 3 | 7 | 0 | 4 | 0 | 12 | 0 | 3 | 3
Not Completed | 0 | 7 | 5 | 5 | 2 | 6 | 2 | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5: Dose escalation with rebastinib 50 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
- Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5: Dose expansion in TNBC participants. Rebastinib 50 mg BID PO in 21-day cycles in combination with carboplatin administered by IV infusion at AUC5 at Day 1 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Total
Number analyzed (Participants) | 3 | 14 | 5 | 9 | 2 | 18 | 2 | 6 | 11 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 4 | 7 | 2 | 9 | 2 | 2 | 5 | 43
  >=65 years | 0 | 5 | 1 | 2 | 0 | 9 | 0 | 4 | 6 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 4 | 9 | 2 | 18 | 2 | 2 | 5 | 53
  Male | 0 | 6 | 1 | 0 | 0 | 0 | 0 | 4 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 8
  Not Hispanic or Latino | 1 | 11 | 5 | 9 | 1 | 18 | 2 | 6 | 8 | 61
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  White | 3 | 13 | 5 | 8 | 1 | 17 | 2 | 6 | 10 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 14 | 5 | 9 | 2 | 18 | 2 | 6 | 11 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants who experienced serious adverse events (SAE) and adverse events (AE).
Time Frame: Baseline up to 2.32 years
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Number analyzed (Participants) | 3 | 14 | 5 | 9 | 2 | 18 | 2 | 6 | 11
Participants
  Any SAE | 2 | 4 | 1 | 5 | 0 | 6 | 0 | 2 | 6
  Any AE | 3 | 13 | 5 | 9 | 2 | 18 | 2 | 6 | 11

2. Primary Outcome: Objective Response Rate (ORR) (Dose Expansion Phase)
Description: Percentage of participants who achieved an objective response of Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumor (RECIST) v1.1. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Time from CR or PR to disease progression or death due to any cause (Up to 1.53 years)
Population: Expansion Phase mITT participants that were evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Number analyzed (Participants) | 9 | 2 | 18 | 2 | 6 | 11
percentage of participants | 0 [0.0 to 28.3] | 0 [0.0 to 77.6] | 16.7 [4.7 to 37.7] | 100 [22.4 to 100.0] | 0 [0.0 to 39.3] | 0 [0.0 to 23.8]

3. Secondary Outcome: Objective Response Rate (ORR) (Dose Escalation Phase)
Description: as for outcome 2
Time Frame: Time from CR or PR to disease progression or death due to any cause (Up to 1.53 years)
Population: Escalation Phase mITT participants that were evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6
Number analyzed (Participants) | 3 | 12 | 5
percentage of participants | 0 [0.0 to 63.2] | 0 [0.0 to 22.1] | 0 [0.0 to 45.1]

4. Secondary Outcome: Duration of Response (DOR)
Description: Time from first partial response (PR) or complete response (CR) to disease progression (PD) or death due to any cause. Evaluation of radiographic disease assessment per Response Evaluation Criteria in Solid Tumor (RECIST v1.1). CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Time from PR or CR to PD or Death due to Any Cause (up to 1.53 years)
Population: mITT participants that had CR or PR and were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
months |  |  |  |  |  | 11.8 [NA to NA] — The 90% Confidence Interval (CI) was not estimable due to insufficient number of events. | 13.5 [8.6 to NA] — The 90% CI was not estimable due to insufficient number of events. |  |

5. Secondary Outcome: Time to Progression (TTP)
Description: Time from first dose of study drug to the first documentation of progressive disease (PD). Participants were considered to have progressive disease if they had documented progression based on radiologic assessment according to RECIST v1.1. RECIST v1.1 defined disease progression as at least a 20% increase in the sum of the disease measurements for measurable lesions, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions.
Time Frame: First Dose of Study Drug to PD (Up to 1.63 years)
Population: mITT participants that were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Number analyzed (Participants) | 2 | 6 | 4 | 7 | 2 | 11 | 2 | 2 | 6
months | 1.4 [0.9 to NA] — The 90% CI was not estimable due to insufficient number of events. | 4.0 [1.4 to NA] — The 90% CI was not estimable due to insufficient number of events. | 2.3 [1.2 to NA] — The 90% CI was not estimable due to insufficient number of events. | 1.5 [1.1 to 3.2] | 1.3 [1.2 to NA] — The 90% CI was not estimable due to insufficient number of events. | 6.7 [4.6 to 13.3] | 14.6 [9.8 to NA] — The 90% CI was not estimable due to insufficient number of events. | NA [4.5 to NA] — TTP median and 90% CI were not estimable due to insufficient number of events. | 4.9 [3.2 to NA] — The 90% CI was not estimable due to insufficient number of events.

6. Secondary Outcome: Progression-free-survival (PFS)
Description: Time from first dose of study drug to disease progression (PD) or death due to any cause. Participants who undergo surgical resection of target or non-target lesions, who have received other anticancer treatments, including surgical resection or radiation (other than palliative radiation to pre-existing bone metastases'), or who do not have a documented date of progression or death due to any cause will be censored at the date of the last assessment. Disease progression per RECIST v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: First Dose of Study Drug to PD or Death due to Any Cause (up to 1.63 years)
Population: mITT participants that were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Number analyzed (Participants) | 3 | 12 | 5 | 9 | 2 | 18 | 2 | 6 | 11
months | 1.4 [0.9 to NA] — The 90% CI was not estimable due to insufficient number of events. | 4.0 [1.4 to NA] — The 90% CI was not estimable due to insufficient number of events. | 2.3 [1.2 to NA] — The 90% CI was not estimable due to insufficient number of events. | 1.5 [1.1 to 3.2] | 1.3 [1.2 to NA] — The 90% CI was not estimable due to insufficient number of events. | 6.7 [4.6 to 13.3] | 14.6 [9.8 to NA] — The 90% CI was not estimable due to insufficient number of events. | NA [4.5 to NA] — PFS median and 90% CI were not estimable due to insufficient number of events. | 4.8 [3.2 to 6.5]

7. Secondary Outcome: Overall Survival (OS)
Description: Time from baseline C1 D1 to date of death due to any cause. Participants who are still alive or who are lost to follow-up will be censored at the date of last contact.
Time Frame: Baseline to death due to any cause (Up to 2.12 years)
Population: mITT participants that were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
Number analyzed (Participants) | 3 | 12 | 5 | 9 | 2 | 18 | 2 | 6 | 11
months | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [1.8 to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | NA [NA to NA] — OS median and 90% CI were not estimable due to insufficient number of events. | 9.9 [4.0 to NA] — The 90% CI was not estimable due to insufficient number of events.

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Rebastinib (Part 1)
Description: Cmax of rebastinib
Time Frame: Part 1: Cycle (C) 1 Day (D) 1, C2 D1 (Cycle = 21 Days)
Population: Part 1 participants who received any study drug and had evaluable Cmax data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6
Number analyzed (Participants) | 3 | 13 | 3
Nanograms per milliliter (ng/mL)
  C1 D1 | 92.2 (157) | 120 (106) | 144 (103)
  C2 D1: number analyzed (Participants) | 3 | 8 | 3
  C2 D1 | 190 (106) | 151 (67.8) | 323 (18.2)

9. Secondary Outcome: PK: Area Under the Concentration-time Curve 0-3 Hours (AUC 0-3 Hours) (Part 1)
Description: Measure the AUC 0-3 hours
Time Frame: Part 1: Cycle (C) 1 Day (D) 1, C2 D1 (Cycle = 21 Days)
Population: Part 1 participants who received any study drug and had evaluable AUC data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms hour per milliliter (ng*h/mL)
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6
Number analyzed (Participants) | 3 | 13 | 3
Nanograms hour per milliliter (ng*h/mL)
  C1 D1 | 186 (153) | 150 (125) | 230 (116)
  C2 D1: number analyzed (Participants) | 3 | 8 | 3
  C2 D1 | 380 (88.3) | 262 (103) | 369 (98.7)

ADVERSE EVENTS:
Time Frame: Baseline up to 2.32 years
Arm/Group | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/14 | 1/5 | 0/9 | 0/2 | 0/18 | 0/2 | 0/6 | 3/11
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/14 | 1/5 | 5/9 | 0/2 | 6/18 | 0/2 | 2/6 | 6/11
Other Adverse Events (participants affected / at risk) | 3/3 | 13/14 | 5/5 | 9/9 | 2/2 | 18/18 | 2/2 | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 (N=3) | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 (N=14) | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 (N=5) | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 (N=9) | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 (N=2) | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 (N=18) | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 (N=2) | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 (N=6) | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5 (N=11)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort 1 Escalation Rebastinib 50 mg + Carboplatin AUC5 (N=3) | Part 1 Cohort 2 Escalation Rebastinib 100 mg + Carboplatin AUC5 (N=14) | Part 1 Cohort 3 Escalation Rebastinib 100 mg + Carboplatin AUC6 (N=5) | Part 2 Cohort 1 Expansion Rebastinib 50 mg + Carboplatin AUC5 (N=9) | Part 2 Cohort 1 Expansion Rebastinib 100 mg + Carboplatin AUC5 (N=2) | Part 2 Cohort 2 Expansion Rebastinib 50 mg + Carboplatin AUC5 (N=18) | Part 2 Cohort 2 Expansion Rebastinib 100 mg + Carboplatin AUC5 (N=2) | Part 2 Cohort 3 Expansion Rebastinib 50 mg + Carboplatin AUC5 (N=6) | Part 2 Cohort 3 Expansion Rebastinib 100 mg + Carboplatin AUC5 (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (3) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 2 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 5 (9) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Refraction disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 9 (11) | 1 (1) | 4 (5) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (8) | 1 (1) | 0 (0) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 7 (9) | 1 (1) | 2 (2) | 6 (6)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 2 (2) | 5 (6)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (5) | 2 (3) | 6 (6) | 0 (0) | 11 (17) | 2 (3) | 1 (1) | 5 (7)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (5) | 1 (1) | 1 (2) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Blood lactate dehydrogenase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 1 (1) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (5) | 0 (0) | 9 (34) | 1 (2) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (4) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 2 (3) | 1 (1) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (7) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Trial terminated on May 23, 2022, due to development program termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT03717415/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT03717415/SAP_001.pdf